CLINICAL TRIAL: NCT02397889
Title: Randomized Controlled Trial of Repeated-Dose Intravenous Ketamine for PTSD
Brief Title: Ketamine as a Treatment for Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Adriana Feder, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 15-0265
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: posttraumatic stress disorder; PTSD; ketamine; trauma; treatment; New York; NYC
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental ketamine group (Experimental): This arm will receive 0.5mg/kg repeated dose ketamine (6 infusions, 3 per week for 2 weeks).
  Interventions: Drug: Ketamine
- Active control midazolam group (Active Comparator): This arm will receive 0.045mg/kg repeated dose midazolam (6 infusions, 3 per week for 2 weeks).
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — This arm will receive 0.5mg/kg repeated dose ketamine (6 intravenous infusions, 3 per week for 2 weeks).
  Other Names: Generic only
  Arms: Experimental ketamine group
Drug: Midazolam — This arm will receive 0.045mg/kg repeated dose intravenous midazolam (6 intravenous infusions, 3 per week for 2 weeks).
  Other Names: Generic only
  Arms: Active control midazolam group

SUMMARY:
The purpose of this study is to study new ways to treat post-traumatic stress disorder (PTSD). Current treatments for PTSD do not work for everyone and it can take time to determine whether a person responds to a chosen treatment. The purpose of this study is to see whether ketamine, when given repeatedly intravenously can produce a quick and persistent improvement in PTSD symptoms. At higher doses, ketamine has been used for many years as an anesthetic for medical procedures, and at lower doses may be an effective treatment in patients with major depression and PTSD. Ketamine given for PTSD is investigational, which means that the FDA has not yet approved the drug for treating this condition. In this study, the effects of ketamine will be compared to those of midazolam. Midazolam has similar acute anesthetic effects compared to ketamine but has not been shown to treat or alleviate any symptoms of PTSD. This makes midazolam an appropriate substance to gauge whether ketamine can treat or alleviate PTSD symptoms thereby acting as what we call an active control.

DETAILED DESCRIPTION:
Ketamine is an approved medication in several countries for the induction of general anesthesia and for use as adjunct to other anesthetics. Intravenous ketamine is being developed and tested for the treatment of posttraumatic stress disorder (PTSD).

All subjects will be administered the study medication by the study anesthesiologists and under the direct supervision of the investigator or designee. On all dosing days, all subjects must remain at the clinical site until at least 4 hours post-dose (or longer if required for study procedures) and will be accompanied by a responsible adult when discharged from the clinical site. The end of study will occur when the last subject in the trial completes his/her last study assessment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18-65 years of age;
* Participants must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign a written informed consent document;
* Participants must fulfill DSM-5 criteria for current civilian or combat-related PTSD
* Women must be using a medically accepted reliable means of contraception (if using an oral contraceptive medication, they must also be using a barrier contraceptive) or not be of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year);
* Women of childbearing potential must have a negative pregnancy test at screening and prior to each intravenous infusion;
* Participants must be able to identify a family member, physician, or friend (i.e. someone who knows them well) who will participate in a Treatment Contract (and e.g. contact the study physician on their behalf in case manic symptoms or suicidal thoughts develop).

Exclusion criteria:

* Women who plan to become pregnant, are pregnant or are breast-feeding
* Serious, unstable medical illnesses such as hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease, including gastro-esophageal reflux disease, obstructive sleep apnea, history of difficulty with airway management during previous anesthetics, ischemic heart disease and uncontrolled hypertension, and history of severe head injury;
* Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
* Renal impairment, as reflected by a BUN >20 mg/dL, and/or creatinin clearance of >1.3 mg/dL;
* Thyroid impairment, as reflected by TSH> 4.2 mU/L Patients with uncorrected hypothyroidism or hyperthyroidism;
* Hormonal treatment (e.g., estrogen) started in the 3 months prior to the first infusion day;
* Use of evidence-based individual psychotherapy (such as prolonged exposure) during the study;
* History of autism, mental retardation, pervasive developmental disorders, or Tourette's syndrome; History of one or more seizures without a clear and resolved etiology;
* History of (hypo)mania;
* Past or current presence of psychotic symptoms, or diagnosis of a lifetime psychotic disorder including schizophrenia or schizoaffective disorder;
* Drug or alcohol abuse or dependence within the preceding 3 months
* Previous recreational use of ketamine or PCP;
* Current diagnosis of bulimia nervosa or anorexia nervosa;
* Diagnosis of schizotypal or antisocial personality disorder
* Patients judged clinically to be at serious and imminent suicidal or homicidal risk.
* A blood pressure of one reading over 160/90 or two separate readings over 140/90 at screen or baseline visits
* Patients who report current treatment with a benzodiazepine, an opioid medication, or a mood stabilizer (such as valproic acid or lithium) within 2 weeks prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05-18; Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Feder, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Depression and Anxiety Center (DAC), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feder A, Costi S, Rutter SB, Collins AB, Govindarajulu U, Jha MK, Horn SR, Kautz M, Corniquel M, Collins KA, Bevilacqua L, Glasgow AM, Brallier J, Pietrzak RH, Murrough JW, Charney DS. A Randomized Controlled Trial of Repeated Ketamine Administration for Chronic Posttraumatic Stress Disorder. Am J Psychiatry. 2021 Feb 1;178(2):193-202. doi: 10.1176/appi.ajp.2020.20050596. Epub 2021 Jan 5. PMID 33397139

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Ketamine Group: 0.5mg/kg repeated dose ketamine (6 infusions, 3 per week for 2 weeks).
- Active Control Midazolam Group: 0.045mg/kg repeated dose midazolam (6 infusions, 3 per week for 2 weeks).
Period: Overall Study
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (13.8) | 38.5 (13.0) | 38.9 (13.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females | 13 | 10 | 23
  Males | 1 | 5 | 6
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 9 | 7 | 16
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Current treatment with psychotropic medication [Count of Participants; unit: Participants] — Number of participants on current treatment with psychotropic medication
  Participants | 7 | 6 | 13
Clinician Administered PTSD Scale (CAPS-5) score [Mean (Standard Deviation); unit: units on a scale] — Clinician Administered PTSD Scale (CAPS-5) score, past month - full range score from 0-80, with higher scores indicating greater PTSD symptoms
  units on a scale | 41.9 (6.1) | 40.1 (5.9) | 40.9 (5.9)
The Impact of Events Scale - Revised (IES-R) [Mean (Standard Deviation); unit: units on a scale] — The Impact of Events Scale - Revised (IES-R) past 24 hours - full range score from 0-88, with higher scores indicating greater PTSD symptoms
  units on a scale | 41.4 (14.0) | 48.3 (20.1) | 44.8 (17.3)
Montgomery Asberg Depression Rating Scale (MADRS) score [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale (MADRS) score, past week - full range score from 0-60, with higher scores indicating greater depressive symptoms
  units on a scale | 27.9 (6.8) | 26.9 (7.7) | 27.4 (7.2)
Montgomery Asberg Depression Rating Scale (MADRS) score [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale (MADRS) score, past 24 hours
  units on a scale | 26.4 (6.6) | 25.3 (9.0) | 25.8 (7.8)
Duration of PTSD [Mean (Standard Deviation); unit: years] | 15.1 (17.8) | 14.6 (7.8) | 14.9 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
Description: full range score from 0-80, with higher scores indicating greater PTSD symptoms
Time Frame: 2 weeks after the first infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group
Number analyzed (Participants) | 15 | 15
score on a scale | 22.5 (14.4) | 33.2 (11.8)

2. Secondary Outcome: The Impact of Event Scale - Revised (IES-R)
Description: full range score from 0-88, with higher scores indicating greater PTSD symptoms
Time Frame: 24 hours after the first drug infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group
Number analyzed (Participants) | 15 | 15
score on a scale | 19.7 (15.2) | 24.8 (13.1)

3. Secondary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: full range score from 0-60, with higher scores indicating greater depressive symptoms
Time Frame: 24 hours after the first drug infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group
Number analyzed (Participants) | 15 | 15
score on a scale | 16.5 (9.6) | 17.1 (9.4)

4. Secondary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: full range score from 0-60, with higher scores indicating greater depressive symptoms
Time Frame: 2 weeks after the first drug infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group
Number analyzed (Participants) | 15 | 15
score on a scale | 14.7 (12.1) | 21.9 (8.5)

5. Secondary Outcome: Quick Inventory of Depression Symptomatology - Self-Report (QIDS-SR)
Description: full range score from 0-27, with higher scores indicating greater depressive symptoms
Time Frame: 2 weeks after the first drug infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group
Number analyzed (Participants) | 15 | 15
score on a scale | 6.6 (7.1) | 6.7 (5.4)

6. Secondary Outcome: Number of Participants With Patient-Rated Inventory of Side Effects (PRISE)
Description: All side effects listed in Adverse Event section.
Time Frame: up to 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

ADVERSE EVENTS:
Time Frame: up to 21 weeks
Arm/Group | Experimental Ketamine Group | Active Control Midazolam Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Ketamine Group (N=15) | Active Control Midazolam Group (N=15)
Diarrhea (Gastrointestinal disorders) | 3 | 4
Dry mouth (Gastrointestinal disorders) | 2 | 0
Nausea/Vomiting (Gastrointestinal disorders) | 7 | 6
Palpitation (Cardiac disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Increased persipiration (Skin and subcutaneous tissue disorders) | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 6
Tremors (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 6 | 2
Blurred vision (Eye disorders) | 10 | 0
Difficulty urinating (Renal and urinary disorders) | 1 | 1
Painful urination (Renal and urinary disorders) | 0 | 1
Frequent urination (Renal and urinary disorders) | 1 | 0
Difficulty sleeping (General disorders) | 2 | 0
Sleeping too much (General disorders) | 1 | 0
Loss of sexual desire (Reproductive system and breast disorders) | 1 | 0
Trouble achieving orgasm (Reproductive system and breast disorders) | 1 | 0
Anxiety (General disorders) | 1 | 0
Poor concentration (General disorders) | 4 | 1
Fatigue (General disorders) | 7 | 14
Decreased energy (General disorders) | 1 | 1
Other (General disorders) | 15 | 10

LIMITATIONS AND CAVEATS:
Exclusion of patients with comorbid psychotic, bipolar, or current alcohol or substance use disorders to protect against worsening of psychotic symptoms or abuse potential, which may limit generalizability of our findings to individuals with PTSD and these comorbid disorders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT02397889/Prot_SAP_000.pdf